CLINICAL TRIAL: NCT06093854
Title: The Efficacy and Safety of Intraoperative Radiotherapy Vesus Stereotactic Body Radiotherapy in Managing Spinal Metastases: A Prospective, Single-center, Open-label, Non-inferior, Randomized Controlled Trial
Brief Title: Intraoperative Radiotherapy in Treating Spinal Metastases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Haifeng Wei, MD, PhD, Professor, Chief Surgeon, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022SL052
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Spinal Metastases
Keywords: spinal metastases; intraoperative radiotherapy; stereotactic body radiotherapy; decompression surgery
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: 1. Decompression surgery + IORT (15-20 Gy, 20-50min）
  2. Decomression surgery + postoperative SBRT ( 30Gy, 5 fractions, 3 weeks)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompression surgery + IORT (Experimental): Decompression surgery + IORT (15-20 Gy, 20-50min）
  Interventions: Radiation: Intraoperative radiotherapy (IORT)
- Decompression surgery + postoperative SBRT (Active Comparator): Decompression surgery + postoperative SBRT (30Gy, 5 fractions, 3 weeks)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Intraoperative radiotherapy (IORT) — Intraoperative radiotherapy (IORT, 15-20 Gy, 20-50min)
  Arms: Decompression surgery + IORT
Radiation: Stereotactic body radiotherapy (SBRT) — postoperative stereotactic body radiotherapy (SBRT, 30Gy, 5 fractions, 3 weeks)
  Arms: Decompression surgery + postoperative SBRT

SUMMARY:
In order to provide theoretical evidence for the comprehensive and standardized treatment of spinal metastases with pathological fractures and/or spinal cord compression, the investigators conduct this trial to investigate the efficacy and safety of IORT and postoperative SBRT in adjuvant treatment of metastatic spinal tumors after posterior decompression surgery by recruiting patients with spinal metastases who met the inclusion criteria, and randomly divided them into the following treatment cohorts: 1) decompression surgery + IORT (15-20 Gy, 20-50min）; 2) decompression surgery and postoperative SBRT(30Gy, 5 fractions, 3 weeks).

DETAILED DESCRIPTION:
Spine is the most common metastatic site for advanced malignancies, accounting for about 70% of all patients with bone metastasis. Approximately 40% -70% of patients with advanced cancer eventually develop spinal metastases.

Spinal metastases require multidisciplinary treatments, and surgical decompression surgery is the preferred treatment in managing spinal metastases with bone related events, especially those with spinal cord compression. The purpose of decompression surgery is to directly relieve nerve compression, alleviate pain, rebuild spinal stability, and reduce tumor burden, which improves the quality of life, and extend the life span indirectly.

At the same time, radiotherapy is also an indispensable treatment for spinal metastases after surgical decompression. The purpose of radiotherapy is to remove residual tumor lesions, alleviate pain, and prevent further pathological fractures. Recent years have witnessed the rapid development of stereotactic bone radiotherapy (SBRT). As reported, SBRT can not only increase the radiation dose at the tumor site, but also reduce radiation damage to the spinal cord and surrounding normal tissues, which is the preferred adjuvant treatment for patients with metastatic spinal tumors. However, SBRT has the several risks, including radiation myelitis, delayed vertebral pathological fractures, local skin allergies, radiotherapy side effects in the esophagus and lungs, and duodenal perforation. Moreover, stereotactic radiotherapy technology has higher costs compared to traditional external beam radiotherapy.

Recently, the application of intraoperative radiotherapy (IORT) can effectively reduce the direct radiation for surrounding normal tissues and maximally eliminate the residual tumor cells. The advantages of IORT include: ① immediate reduction of the possibility of tumor cell expansion after surgery; ② Safe direct radiation and effective protection of normal tissues beyond the radiation depth; ③ To effectively protect adjacent normal tissues, light-limiting tubes with different diameters can be selected based on the size and range of tumor; ④ Shortening treatment course with lower costs and better compliance; ⑤ Slight systemic side effects and bone marrow suppression.

To the knowledge, no research focuses on the efficacy of IORT and SBRT in the adjuvant treatment of spinal metastases. Therefore, in order to provide theoretical evidence for the comprehensive and standardized treatment of spinal metastases with pathological fractures and/or spinal cord compression, the investigators conduct this trial to investigate the efficacy and safety of IORT and postoperative SBRT in adjuvant treatment of metastatic spinal tumors after posterior decompression surgery by recruiting patients with spinal metastases who met the inclusion criteria, and randomly divided them into the following treatment cohorts: 1) decompression surgery + IORT (15-20 Gy, 20-50min）; 2) decompression surgery and postoperative SBRT(30Gy, 5 fractions, 3 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spinal metastases;
* Estimated survival time more than 3 months;
* The spinal instability neoplastic score (SINS) >12;
* The general condition allows to recieve surgery;
* Single or multiple metastatic lesions with only one site presenting epidural spinal cord compression;
* signed informed consent.

Exclusion Criteria:

* Clinical diagnosis of primary spinal tumors;
* Presence of metastases in central nerve system;
* Isolated lesion undergoing en bloc resection;
* Mental disorder and/or intellectual dificiency;
* Refusing to accept follow-up;
* without signing informed consent.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 2 years
  The local control of tumor in the surgical field

SECONDARY OUTCOMES:
Health-related quality of life | 2 years
  The "Functional Assessment of Cancer Therapy -General" (FACT-G) Scale (Minimum: 0; Maximum: 108 ) is utilized to evaluate the health-related quality of life after treatments, and higher scores mean a worse outcome.
Progression-free survival | 2 years
  The survival time between the day after treatments and the date of any evidence proving tumor progression or final follow-up
Overall survival | 2 years
  The survival time between the day after treatments and the date of all-cause death or final follow-up
Radiation-related complications | 2 years
  The complications assciated with the radiation process

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barzilai O, Laufer I, Yamada Y, Higginson DS, Schmitt AM, Lis E, Bilsky MH. Integrating Evidence-Based Medicine for Treatment of Spinal Metastases Into a Decision Framework: Neurologic, Oncologic, Mechanicals Stability, and Systemic Disease. J Clin Oncol. 2017 Jul 20;35(21):2419-2427. doi: 10.1200/JCO.2017.72.7362. Epub 2017 Jun 22. PMID 28640703
- [Background] Laufer I, Rubin DG, Lis E, Cox BW, Stubblefield MD, Yamada Y, Bilsky MH. The NOMS framework: approach to the treatment of spinal metastatic tumors. Oncologist. 2013 Jun;18(6):744-51. doi: 10.1634/theoncologist.2012-0293. Epub 2013 May 24. PMID 23709750
- [Background] Calvo FA. Intraoperative irradiation: precision medicine for quality cancer control promotion. Radiat Oncol. 2017 Feb 2;12(1):36. doi: 10.1186/s13014-017-0764-5. PMID 28148287
- [Background] Vaidya JS, Bulsara M, Baum M, Alvarado M, Bernstein M, Massarut S, Saunders C, Sperk E, Wenz F, Tobias JS; TARGIT-A investigators. Intraoperative radiotherapy for breast cancer: powerful evidence to change practice. Nat Rev Clin Oncol. 2021 Mar;18(3):187-188. doi: 10.1038/s41571-021-00471-7. No abstract available. PMID 33495552
- [Result] Barzilai O, McLaughlin L, Amato MK, Reiner AS, Ogilvie SQ, Lis E, Yamada Y, Bilsky MH, Laufer I. Predictors of quality of life improvement after surgery for metastatic tumors of the spine: prospective cohort study. Spine J. 2018 Jul;18(7):1109-1115. doi: 10.1016/j.spinee.2017.10.070. Epub 2017 Nov 6. PMID 29122701
- [Result] Patchell RA, Tibbs PA, Regine WF, Payne R, Saris S, Kryscio RJ, Mohiuddin M, Young B. Direct decompressive surgical resection in the treatment of spinal cord compression caused by metastatic cancer: a randomised trial. Lancet. 2005 Aug 20-26;366(9486):643-8. doi: 10.1016/S0140-6736(05)66954-1. PMID 16112300
- [Result] Correia D, Moullet B, Cullmann J, Heiss R, Ermis E, Aebersold DM, Hemmatazad H. Response assessment after stereotactic body radiation therapy for spine and non-spine bone metastases: results from a single institutional study. Radiat Oncol. 2022 Feb 21;17(1):37. doi: 10.1186/s13014-022-02004-7. PMID 35189919
- [Result] Thibault I, Chang EL, Sheehan J, Ahluwalia MS, Guckenberger M, Sohn MJ, Ryu S, Foote M, Lo SS, Muacevic A, Soltys SG, Chao S, Gerszten P, Lis E, Yu E, Bilsky M, Fisher C, Schiff D, Fehlings MG, Ma L, Chang S, Chow E, Parelukar WR, Vogelbaum MA, Sahgal A. Response assessment after stereotactic body radiotherapy for spinal metastasis: a report from the SPIne response assessment in Neuro-Oncology (SPINO) group. Lancet Oncol. 2015 Dec;16(16):e595-603. doi: 10.1016/S1470-2045(15)00166-7. PMID 26678212
- [Result] Sahgal A, Myrehaug SD, Siva S, Masucci GL, Maralani PJ, Brundage M, Butler J, Chow E, Fehlings MG, Foote M, Gabos Z, Greenspoon J, Kerba M, Lee Y, Liu M, Liu SK, Thibault I, Wong RK, Hum M, Ding K, Parulekar WR; trial investigators. Stereotactic body radiotherapy versus conventional external beam radiotherapy in patients with painful spinal metastases: an open-label, multicentre, randomised, controlled, phase 2/3 trial. Lancet Oncol. 2021 Jul;22(7):1023-1033. doi: 10.1016/S1470-2045(21)00196-0. Epub 2021 Jun 11. PMID 34126044
- [Result] Myrehaug S, Sahgal A, Hayashi M, Levivier M, Ma L, Martinez R, Paddick I, Regis J, Ryu S, Slotman B, De Salles A. Reirradiation spine stereotactic body radiation therapy for spinal metastases: systematic review. J Neurosurg Spine. 2017 Oct;27(4):428-435. doi: 10.3171/2017.2.SPINE16976. Epub 2017 Jul 14. PMID 28708043
- [Result] Orecchia R, Veronesi U, Maisonneuve P, Galimberti VE, Lazzari R, Veronesi P, Jereczek-Fossa BA, Cattani F, Sangalli C, Luini A, Caldarella P, Venturino M, Sances D, Zurrida S, Viale G, Leonardi MC, Intra M. Intraoperative irradiation for early breast cancer (ELIOT): long-term recurrence and survival outcomes from a single-centre, randomised, phase 3 equivalence trial. Lancet Oncol. 2021 May;22(5):597-608. doi: 10.1016/S1470-2045(21)00080-2. Epub 2021 Apr 9. PMID 33845035
- [Result] Vaidya JS, Bulsara M, Saunders C, Flyger H, Tobias JS, Corica T, Massarut S, Wenz F, Pigorsch S, Alvarado M, Douek M, Eiermann W, Brew-Graves C, Williams N, Potyka I, Roberts N, Bernstein M, Brown D, Sperk E, Laws S, Sutterlin M, Lundgren S, Holmes D, Vinante L, Bozza F, Pazos M, Le Blanc-Onfroy M, Gruber G, Polkowski W, Dedes KJ, Niewald M, Blohmer J, McCready D, Hoefer R, Kelemen P, Petralia G, Falzon M, Baum M, Joseph D. Effect of Delayed Targeted Intraoperative Radiotherapy vs Whole-Breast Radiotherapy on Local Recurrence and Survival: Long-term Results From the TARGIT-A Randomized Clinical Trial in Early Breast Cancer. JAMA Oncol. 2020 Jul 1;6(7):e200249. doi: 10.1001/jamaoncol.2020.0249. Epub 2020 Jul 9. PMID 32239210
- [Result] Wenz F, Schneider F, Neumaier C, Kraus-Tiefenbacher U, Reis T, Schmidt R, Obertacke U. Kypho-IORT--a novel approach of intraoperative radiotherapy during kyphoplasty for vertebral metastases. Radiat Oncol. 2010 Feb 11;5:11. doi: 10.1186/1748-717X-5-11. PMID 20149237
- [Result] Bludau F, Welzel G, Reis T, Schneider F, Sperk E, Neumaier C, Ehmann M, Clausen S, Obertacke U, Wenz F, Giordano FA. Phase I/II trial of combined kyphoplasty and intraoperative radiotherapy in spinal metastases. Spine J. 2018 May;18(5):776-781. doi: 10.1016/j.spinee.2017.09.011. Epub 2017 Sep 28. PMID 28962909